CLINICAL TRIAL: NCT06364501
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Anti-tumor Activity of KH801 Injection in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Trial of KH801
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Kanghong Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KH801
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): KH801 will be sequentially escalated at the dose of 0.01 mg/kg, 0.1 mg/kg, 0.3 mg/kg, 1.0 mg/kg , 3.0 mg/kg, 6.0 mg/kg , 10.0 mg/kg, administered via intravenous infusion every 2 weeks in 28-day treatment cycles.
  Interventions: Drug: KH801

INTERVENTIONS:
Drug: KH801 — KH801 is an injection solution

SUMMARY:
KH801 is a injection used for advanced solid tumors which must be diluted with 5% Dextrose Or 0.9% sodium chloride Injection.

This study is expected to include a total of approximately 17-42 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent voluntarily.
2. Age ≥ 18 years old (subject to the date of signing the informed consent form), both genders.
3. With an expected life expectancy of ≥ 3 months.
4. With an ECOG（Eastern Cooperative Oncology Group Performance Status） performance status score of 0-1.
5. Patients with locally advanced unresectable or metastatic malignant solid tumors confirmed by histology, (including but not limited to breast cancer, lung cancer, ovarian cancer, colorectal cancer and other solid tumors) who failed or unable to tolerate previous standard treatments.
6. With at least one measurable target lesion was evaluated according to RECIST v1.1 criteria. Measurable target lesions were defined as non-lymph node lesions with the longest single diameter ≥ 10mm, or lymph node lesions with a short diameter ≥ 15mm.
7. The organ function reserve of patients before enrollment should meet the following laboratory test values:

   7.1 Hematology: Neutrophil count ≥ 1.5 × 109/L, hemoglobin ≥ 90g/L, platelets ≥ 100 × 109/L ( Use of hematopoietic growth factor drugs within the first two weeks of screening is not allowed to improve the detection value and meet inclusion criteria); 7.2 Liver function: Total bilirubin ≤ 1.5 x ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN (if there is liver metastasis or hepatocellular carcinoma(HCC), ALT and AST ≤ 5 x ULN); 7.3 Renal function: serum creatinine ≤ 1.5 × ULN, or creatinine clearance rate ≥ 50 milliliter（mL)/min (calculated using Cockcroft Gault formula, see Appendix 5 for details); Urinary protein<2+, or urinary protein ≥ 2+and 24-hour urine protein quantification<1g; 7.4 Coagulation function: prothrombin time (PT), international normalized ratio (INR), and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN (except for patients receiving anticoagulant therapy).
8. Female patients with fertility or male patients with partners with fertility must start using efficient contraceptive measures 7 days before the first dose and continue until 6 months after the last dose (excluding those who have undergone sterilization surgery (such as bilateral tubal ligation, oophorectomy, or hysterectomy). Female patients with fertility must have a negative blood pregnancy test within 7 days before the first administration.
9. Patients must recover from acute toxic reactions caused by previous anti-tumor treatments (CTCAE ≤ level 1), except for the following situations: a. hair loss; b. Skin pigmentation; c. Grade 2 ande below neurotoxicity; d. The long-term toxicity caused by radiotherapy cannot be restored according to the judgment of the researchers.

Exclusion Criteria:

1. Patients with primary central nervous system tumors and central nervous system (CNS) metastases (except for patients who have been clinically stable for ≥ 4 weeks after previous surgery or radiotherapy and have discontinued corticosteroid treatment).
2. Patients with interstitial lung disease (ILD) (excluding local interstitial pneumonia caused by radiotherapy), severe chronic obstructive pulmonary disease, and severe pulmonary insufficiency.
3. Positive for human immunodeficiency virus antibody (HIVAb), active hepatitis B virus infection (HBV-DNA copy number ≥ ULN) or active hepatitis C virus infection (HCV-RNA ≥ ULN), as well as other severe active infections that have not been controlled or require treatment.
4. Individuals who have previously received cluster of differentiation 24(CD24) targeted therapy.
5. Previous history of receiving allogeneic hematopoietic stem cell transplantation or other organ transplantation;
6. Patients who have received any anti-tumor treatment (including chemotherapy, hormone therapy, radiotherapy, immunotherapy, or biological therapy) within 4 weeks or 5 half lives of drugs previously used (whichever is longer) before the first dose.
7. Participated in other clinical trials within 4 weeks prior to the first administration.
8. Female subjects in lactation or pregnancy.
9. Previous or current mental/neurological disorders are not limited to schizophrenia, delusions, phobias, obsessive-compulsive disorder, Alzheimer's disease, behavioral and volitional disorders, postpartum mental disorders, paranoid mental disorders, and various organic disorders accompanied by mental disorders.
10. Active autoimmune diseases within the past 2 years (excluding vitiligo, Graves disease, Hashimoto's thyroiditis, or psoriasis that do not require systemic treatment).
11. Have suffered from other malignant tumors within the past 5 years, except for the following situations:

    11.1 Cured non melanoma skin malignant tumors; 11.2 Cervical carcinoma in situ; 11.3 Cured stage I endometrial cancer; 11.4 Curative breast ductal carcinoma in situ or lobular carcinoma in situ, and currently not receiving any systemic treatment; 11.5 Localized prostate cancer, papillary thyroid cancer, or follicular thyroid cancer that has undergone radical surgery and is currently considered cured/long-term stable.
12. Accompanied by active cardiovascular and cerebrovascular diseases:

    12.1 Has experienced myocardial infarction, stroke, bypass surgery, or stent placement within 6 months prior to the first administration; 12.2 Congestive heart failure New York Heart Association(NYHA) III-IV; 12.3 Left ventricular ejection fraction (LVEF)<50%; 12.4 Corrected QT interval(QTC) was prolonged (female>470ms, male>450ms); 12.5 Unstable angina that cannot be controlled by medication, severe arrhythmias that require medication treatment (excluding atrial fibrillation or paroxysmal supraventricular tachycardia); 12.6 Hypertension (systolic blood pressure ≥ 160 millimeters of mercury (mmHg) or diastolic blood pressure ≥ 100mmHg) that cannot be controlled after standardized drug treatment, as well as a history of hypertensive crisis or hypertensive encephalopathy; 12.7 Suffering from major vascular diseases (such as aortic aneurysm, aortic dissection).
13. Patients with deep vein thrombosis (except for those with stable intermuscular vein thrombosis or infusion port thrombosis assessed by the investigators), pulmonary embolism or other serious thromboembolism, or patients with deep vein thrombosis, pulmonary embolism or other serious thromboembolism within 6 months before enrollment, and who are assessed by the investigator to be at risk of recurrence.
14. Patients allergic to immunoglobulin or any component of KH801 injection.
15. Patients who have received live attenuated vaccine within 4 weeks before enrollment or plan to receive live attenuated vaccine during the study period.
16. Patients who have undergone major surgery within 4 weeks before the first dose or plan to have major surgery during the study period.
17. Patients who have any other conditions that render them inappropriate for inclusion in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
MTD | up to 4 weeks
  Maximum tolerated dose (MTD)
DLT | up to 4 weeks
  Dose limiting toxicity (DLT)
RP2D | up to 1 year
  Recommended phase II dose (RP2D)

SECONDARY OUTCOMES:
AE | 30 days after EOT,up to 1 year
  Adverse events
Cmax | up to 12 weeks
  Maximum serum concentration (Cmax) of KH801 will be investigated
Tmax | up to 12 weeks
  Time to maximum serum concentration(Tmax) of KH801 will be investigated
T1/2 | up to 12 weeks
  Half-life (T1/2) of KH801 will be investigated
AUC0-t | up to 12 weeks
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration
CL | up to 12 weeks
  Plasma clearance rate (Cl) is defined the volume of plasma per unit time in which drugs are completely eliminated.
AUC0-inf | up to 12 weeks
  AUC0-inf is defined area under the blood drug concentration time curve from 0 to infinity
anti-drug antibody (ADA) | up to 1 years
  The anti-drug antibody of KH801

OTHER OUTCOMES:
Objective Response Rate（ORR） | through study completion, an average of 1 year
  Objective Response Rate（ORR）is defined as the percentage of participants, who has a complete response (CR) (disappearance of all target lesions) or partial response (PR) (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1
Disease Control Rate (DCR) | through study completion, an average of 1 year
  The Disease Control Rate (DCR) is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD): at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | through study completion, an average of 1 year
  The Duration of Response (DOR) for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Median Progression-Free Survival (mPFS) | through study completion, an average of 1 year
  Median progression free survival (mPFS) refers to the progression free survival that 50% of assessable patients can achieve
Overall Survival（OS) | through study completion, an average of 1 year
  The overall survival period refers to the time period from the start of treatment in a patient's study (whether randomized or single arm trial) until death from any cause

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Central Hospital Affiliated To Shandong First Medical University, Jinan, Shandong
  - West China Second University Hospital,Sichuan University/West China Women's and Children's Hospital, Chengdu, Sichuan